CLINICAL TRIAL: NCT04026880
Title: A Pilot Study To Evaluate The Effect of Testosterone Enanthate On Structural and Functional Characteristics of Pelvic Floor Muscles In Postmenopausal Women With Urinary Incontinence
Brief Title: Testosterone Effects on Pelvic Floor Muscles
Acronym: TPELVIC
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of funds
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Grace Huang, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018P000248
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Urinary Incontinence; Menopause
Keywords: Androgens; Menopause; Urinary Incontinence; Pelvic Floor Muscles
MeSH Terms: conditions — Urinary Incontinence | interventions — testosterone enanthate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Active Comparator): weekly IM administration of 25 mg Testosterone Enanthate for 12 weeks
  Interventions: Drug: Testosterone Enanthate
- Control Arm (Placebo Comparator): Weekly IM administration of placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Testosterone Enanthate — 25 mg testosterone enanthate administered by intramuscular injection weekly for 12 weeks
  Other Names: Delatestryl
  Arms: Treatment Arm
Drug: Placebo — Placebo administered by intramuscular injection weekly for 12 weeks
  Other Names: Inactive comparator
  Arms: Control Arm

SUMMARY:
An proof-of-concept study to determine whether administration of testosterone enanthate weekly results in greater improvements in structural and functional characteristics of pelvic floor muscles and urodynamic parameters in postmenopausal women with urinary incontinence than that associated with placebo administration

DETAILED DESCRIPTION:
Androgen therapy has been widely promoted in women with low serum testosterone levels for the treatment of sexual dysfunction and also for potentially improving body composition, muscle performance, bone mineral density and cognition. Androgens are known to exert direct anabolic effects on skeletal muscle. Testosterone supplementation results in dose-dependent increases in both muscle mass and strength in men. Similarly, our group has also demonstrated that 24-weeks of testosterone administration in hysterectomized women with low testosterone levels was associated with dose and concentration-dependent gains in lean body mass, chest-press power and loaded stair-climb power. Given that androgen receptors have been shown to be expressed throughout the pelvic floor and lower urinary tract, the anabolic effects of androgens on pelvic floor muscles and urethral sphincter may provide a therapeutic option in women with urinary incontinence.

In spite of the recognition of the important role of androgens in regulation of pelvic floor muscle mass and function, no randomized trials of the effects of testosterone or selective androgen receptor modulators have been published. Towards our long-term goal of conducting such a randomized efficacy trial of the effect of androgens in women with urinary incontinence, this initial pilot study will provide important data as a proof-of-the concept that the mass and function of levator ani and other pelvic floor muscles can be increased meaningfully by administration of testosterone, and that the increase in the mass and function of pelvic floor muscles will be associated with significant improvements in urodynamic parameters. Although MRI has been used clinically to evaluate pelvic floor anatomy, dynamic MRI of the pelvic floor muscles coupled with urodynamic studies has not been standardized previously; an important aim of this pilot study is to optimize the procedures for dynamic MR imaging of the pelvic floor structures and couple them with evaluation of urodynamics of the urinary bladder, bladder sphincter, and the urethra. Furthermore, the preliminary estimates of effect size and variance generated in this pilot study will guide the estimates of sample size and statistical power in subsequent larger randomized efficacy trials of androgens in women with urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

1. Medically stable, ambulatory, postmenopausal women, 60 years of age or older
2. A normal mammogram in the preceding 12 months of study entry will be required. Women will be asked to either provide documentation of their last mammogram results or, with their permission, sign a medical release form to allow us to obtain the results of their last mammogram.
3. Able to give informed consent
4. Women with either stress urinary incontinence, or mixed urinary incontinence (stress and urgency)

Exclusion Criteria:

1. Women with endometrial stripe >4 mm on pelvic ultrasound
2. ≥ 1 first-degree relative with breast cancer
3. Previous pelvic surgery (ie. hysterectomy)
4. Women with history of radiation treatment to the pelvis
5. Any neurologic disorder causing urinary incontinence or bladder dysfunction (ie. multiple sclerosis)
6. Estrogen therapy currently or in the past 3 months
7. Women who have been diagnosed with major psychoses or bipolar disorders and/or untreated depression
8. Women with severe depression and/or severe anxiety as measured by the Beck Depression Inventory (BDI-II) and Beck Anxiety Inventory (BAI), respectively
9. Any acute or subacute illness that required hospitalization in the last three months
10. Cancers that require active therapy (not in remission for at least two years) including those with a life expectancy less than 5 years
11. Poorly controlled diabetes mellitus (hemoglobin A1c greater than 8.0%). Subjects on insulin therapy will be excluded.
12. Uncontrolled hypertension defined as an average of two blood pressure readings of greater than 160/100
13. Severe obesity defined as body mass index of greater than 40 kg/m2
14. Current or recent (last 6 months) users of illicit drugs
15. Significant liver function abnormalities, defined as SGOT, SGPT or alkaline phosphatase value of greater than 1.5 times the upper limit of normal or serum bilirubin levels of greater than 1.5 mg/dl will be excluded
16. History of breast, ovarian, or endometrial cancer.
17. History of hyperandrogenic disorders such as moderate to severe hirsutism and/or acne (by self-report), and polycystic ovary disease. Testosterone administration to these patients may exacerbate the underlying disorder.
18. Significant acne, defined as grade 3 on Palatsi Acne Scale
19. Women with a mammogram that requires follow-up every 3-6 months, or those who have any first-degree relatives with breast cancer will be excluded.
20. Women with history of a major cardiovascular event, including angina, congestive heart failure, cerebral vascular accident or history of myocardial infarction or coronary artery angioplasty or bypass surgery
21. Other Medications. Women who have received in the preceding three months drugs known to affect testosterone production or metabolism such as ketoconazole, Megace, anabolic/androgenic steroids for 3 weeks or longer will be excluded. Women taking ≥ 7.5 mg of prednisone or equivalent glucocorticoid dosing will be excluded. We will also exclude women who are taking or have taken in the past three months medications that affect sexual function (e.g., spironolactone, GnRH agonists). Women receiving thyroid hormone replacement therapy may participate in the study if they have been on a stable replacement dose of L-thyroxine for at least six months.
22. Undiagnosed vaginal or vulvar bleeding
23. Women taking concurrent anticoagulants or how have bleeding disorders
24. History of deep vein thrombosis, pulmonary embolism, or other thromboembolic disorder
25. Current enrollment in clinical drug intervention studies in the preceding 90 days
26. Hematocrit < 30% or >48% (Since hematocrit values can transiently increase as a result of dehydration, and the subjects in this trial are required to come after an overnight fast, hematocrit levels may be repeated once if the investigators determine that the initial elevated hematocrit was influenced by dehydration)
27. Women who have previously experienced intolerance to testosterone enanthate injections
28. Unable to undergo MRI of the pelvis (e. g. body containing any metallic medical devices or equipment, including heart pacemakers, metal prostheses, implants or surgical clips, any prior injury from shrapnel or grinding metal, exposure to metallic dusts, metallic shavings or having tattoos containing metallic dyes).

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in pelvic floor muscle volume | 12 weeks
  Pelvic floor muscle volume will be measured by 3-dimensional dynamic pelvic floor magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Change in urine volume at first desire to void | 12 weeks
  Urine volume at first desire to void will be assessed by cystometry
Change in urine volume at first urge to void | 12 weeks
  Urine volume at first urge to void will be assessed by cystometry
Change in maximum cystometric capacity (when the patient feels she can no longer delay micturition) | 12 weeks
  Maximum Cystometric Capacity will be assessed by cystometry
Change in urine flow | 12 weeks
  Rate of urine flow (urine volume voided over time) will be assessed by Uroflowmetry
Change in urethral sphincter contraction strength | 12 weeks
  Strength of urethral sphincter contraction will be assessed by urethral pressure profilometry.
Change in urine leak point pressure | 12 weeks
  Urine leak point pressure will be assessed by cystometry
Change in self-reported urinary incontinence | 12 weeks
  Urinary Incontinence will be assessed by the Urogenital Distress Inventory (UDI-6 Short Form). The UDI-6 Short Form is a questionnaire with 6 questions that assess the presence and severity of urinary incontinence symptoms. Each question has a potential score of 1 to 4. The final UDI-6 score is calculated by adding all scores as explained above, and dividing the result by 6 to obtain a mean value which is in turn multiplied by 25 to obtain the scale score.
  The total scaled score can range from 0 to 100, higher scores indicating more severe urinary incontinence, and lower scores indicating less severe urinary incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Grace Huang, MD, Principal Investigator — Partners Health Care, Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang G, Basaria S, Travison TG, Ho MH, Davda M, Mazer NA, Miciek R, Knapp PE, Zhang A, Collins L, Ursino M, Appleman E, Dzekov C, Stroh H, Ouellette M, Rundell T, Baby M, Bhatia NN, Khorram O, Friedman T, Storer TW, Bhasin S. Testosterone dose-response relationships in hysterectomized women with or without oophorectomy: effects on sexual function, body composition, muscle performance and physical function in a randomized trial. Menopause. 2014 Jun;21(6):612-23. doi: 10.1097/GME.0000000000000093. PMID 24281237